CLINICAL TRIAL: NCT05979376
Title: Efficacy of Dexmedetomidine as an Adjuvant to Quadratus Lumborum Block for Paediatric Groin Surgery:A Randomized Double Blind Study
Brief Title: Efficacy of Dexmedetomidine as an Adjuvant to Quadratus Lumborum Block
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Yagmur Gul, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: E-83045809-604.01.01-631721
Record Dates: First submitted 2023-07-29; First posted 2023-08-07 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Pain, Postoperative
Keywords: dexmedetomidine; bupivacaine; quadratus lumborum block; postoperative pain; regional anesthesia; pediatric anesthesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I (Control group): group I: quadratus lumborum block with 0,25% bupivacaine 0,5 ml/kg
- Group II: groupII: quadratus lumborum block with 0,25%bupivacaine 0,5 ml/kg and dexmedetomidine 0,5 mcg/kg as an adjuvant
- Group III: groupIII: quadratus lumborum block with 0,25% bupivacaine 0,5 ml/kg and dexmedetomidine 1 mcg/kg as an adjuvant

SUMMARY:
This prospective double blinded study will be conducted over 60 pediatric patients ASA (American Association of Anesthesiologists) I and II between the age of 1-7 years old, who will be scheduled for unilateral groin surgery. Patients will be randomly allocated into 3 study groups: Control group that only received local anesthetics ( bupivacaine) Group II bupivacaine with the dexmetedomidine ( 0,5mcg/kg ) and group III bupivacaine with the dexmedetomidine (1mcg/kg).Patients in all groups will receive quadratus lumborum block.

Bradycardia, hypotension, atropine, and bolus fluid infusion requirements will be recorded. When there was up to a 30% decrease in basal mean blood pressure, a crystalloid infusion bolus will be given at 10 ml/kg. When bradycardia occurred , atropine will be given at a dose of 0.02 mg/kg. Patients will be followed up in the postoperative recovery unit for the first 2 hours, and then in the ward. The RAMSEY sedation scale and WATCHA agitation scale were evaluated at 5, 15, 30, and 60 minutes in the postoperative recovery unit. Nausea, vomiting, and other side effects were recorded if present.

Time to first analgesic requirement ( primary outcome) , FLACC Scale scores will be recorded within 24h postoperatively, total dose of analgesic consumption, incidence of postoperative complications as hypotension, bradycardia, vomiting, pruritis and respiratory depression will be recorded.

ELIGIBILITY:
Inclusion Criteria:

The study included children aged 1-7 years with ASA (American Society of Anesthesiologists) I-II, who underwent elective, unilateral, groin surgery (inguinal hernia, orchiopexy, hydrocele) with the consent of their families

Exclusion Criteria:

* Children who were aged outside the range of 1-7 years, with ASA III or higher, allergic to local anesthetics, had an infection in the injection area, had contraindications for regional anesthesia such as coagulopathy, whose families did not give consent, were undergoing laparoscopic orchidopexy, undergoing bilateral surgery, had a body mass index of >30 kg/m2, and were expected to be admitted to the intensive care unit during the postoperative period were excluded from the study

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patient children aged 1-7 years
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
the time to first rescue analgesic requirement | 24 hours
  the time to first rescue analgesic requirement within the first 24 postoperative hours,

SECONDARY OUTCOMES:
postoperative pain scores FLACC (face, legs, activity, cry, and consolability) | 24 hours
  postoperative pain assessment score in children (The scale is scored in a range of 0-10 with 0 representing no pain, 10 representing maximum pain)
additional analgesic consumption | 24 hours
  total analgesic consuption within 24 hours
postoperative sedation scores RAMSEY (Ramsey sedation scale) | 1 hour
  patient's sedation scores within postoperative first one hour (Ramsey sedation score is scored in a range of 1-6 with 1 representing awake; agitated or restless, 6 representing Asleep; no response to glabellar tap or loud auditory stimulus)
incidence of complications | 24 hours
  Incidence of intraoperative and postoperative complications or side effects

CONTACTS AND LOCATIONS:
Overall Officials: PINAR Kendigelen, Prof., Study Director — Istanbul University - Cerrahpasa
Locations (1):
- PINAR Kendigelen, Istanbul, Please Select, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No